CLINICAL TRIAL: NCT03806062
Title: EFFECT OF LOW LEVEL LASER THERAPY VERSUS ELECTROACUPUNCTURE ON POSTNATAL SCANTY MILK SECRETION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48
Record Dates: First submitted 2019-01-13; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Insufficient Lactation
MeSH Terms: conditions — Lactation Disorders | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): 10 mg domperidone 3 times a day after meals) and advice about lactation, nutrition and fluid intake all through the treatment period (4 weeks)
  Interventions: Drug: domperidone
- Laser group (Active Comparator): The laser scan beam was adjusted to the size of the treated breast for 10 minutes with wave length 632.8 nm and power output 25 mw after the end of treatment session on both breasts.
  The mother had one session every other day, three sessions weekly for four weeks. (Total 12 sessions)
  Interventions: Drug: domperidone; Device: He-Ne laser (Bravo TrezaSerie) device
- Electro acupuncture group (Active Comparator): faradic stimulation (Body shaping System, model B-333, made in China) , at the following acupuncture points on both sides: Spleen 6 (Sanyinjiao), Liver 3 (Taichong) and Small Intestine 1 (Shaoze) using surface electrodes
  Interventions: Drug: domperidone; Device: faradic current

INTERVENTIONS:
Drug: domperidone — 10 mg domperidone 3 times a day after meals
Device: He-Ne laser (Bravo TrezaSerie) device — The laser scan beam was adjusted to the size of the treated breast for 10 minutes with wave length 632.8 nm and power output 25 mw after the end of treatment session
  Arms: Laser group
Device: faradic current — faradic stimulation (Body shaping System, model B-333, made in China) , at the following acupuncture points on both sides: Spleen 6 (Sanyinjiao), Liver 3 (Taichong) and Small Intestine 1 (Shaoze)
  Arms: Electro acupuncture group

SUMMARY:
A randomized controlled study conducted on 60 healthy primiparous mothers with insufficient lactation. The participants were divided randomly into three equal groups, Group (A) control, Group (B) received low power He-Ne laser beam on both breasts and Group (C) received faradic current stimulation at Spleen 6, Liver 3 and Small Intestine 1 acupuncture points on both sides, all participants received 10 mg domperidone 3 times a day and advice about lactation, nutrition and fluid intake. Evaluation was done before and after the treatment program

DETAILED DESCRIPTION:
Women in Group (A) acted as a control group and only received medical treatment in the form of 10 mg domperidone 3 times a day after meals) and advice about lactation, nutrition and fluid intake all through the treatment period (4 weeks) Each woman in group (B) lied in supine lying position on the treatment plinth wearing the protective eyewear as precautionary measures for her safety and exposing her breast out of her clothes then the breast was cleaned by alcohol. The laser apparatus was directed perpendicularly over the treated breast at a distance 50 cm from it, all metal objects must be removed from the range of action of laser (i.e. necklaces). The laser scan beam was adjusted to the size of the treated breast for 10 minutes with wave length 632.8 nm and power output 25 mw after the end of treatment session the machine switched off automatically then, it was adjusted again to start irradiation by the same procedures for the other breast. The mother had one session every other day, three sessions weekly for four weeks. (Total 12 sessions). He-Ne laser (Bravo TrezaSerie) device was used. The equipment was designed in compliance with international technical standards UNI EN ISO 9002 and En 46002 and complies with the safety requirements.

Group (B) had received 12 sessions of irradiation by low power He-Ne laser beam on both sides of the breasts 10 minutes on each side. One session every other day, three sessions weekly for four weeks beside the medical treatment (10 mg domperidone 3 times a day after meals) and advice about lactation, nutrition and fluid intake all through the treatment period Group (C) women were treated by faradic stimulation (Body shaping System, model B-333, made in China) , at the following acupuncture points on both sides: Spleen 6 (Sanyinjiao), Liver 3 (Taichong) and Small Intestine 1 (Shaoze) using surface electrodes in addition to medical treatment (10 mg domperidone 3 times a day after meals) and advice about lactation, nutrition and fluid intake allthrough the treatment period

SP-6 Acupuncture Point lies on the inner leg aspect about 3 cm higher than the medial malleolus, along the posterior tibial border. Fig. (2)

LIV-3 Acupuncture Point is the one that lies in the depressed area between the 1st 2 metatarsal bones proximal to the metatarsophalangeal joints on the dorsal foot aspect Fig. (2)

SI.1 Acupuncture point is located on the little finger, ulnar to the distal phalanx, at the intersection of the vertical line of ulnar border of the nail and the horizontal line of the base of the little fingernail. Fig. (2)

Each woman in group (C) was asked to be in a long sitting or half lying position, When the points were located, the electrodes were fastened securely with an adhesive tape or an elastic band to ensure good contact between the skin and the electrode over the acupuncture points. The intensity control of the stimulator was slowly increased until the patient could just feel the stimulation. The session lasted for 30 minutes. One session every other day, 3 sessions weekly for 4 weeks. (Total 12 sessions).

ELIGIBILITY:
Inclusion Criteria:

* Their age ranged between 20 and 35 years old
* 25 to 30 kg/m² body mass index (BMI).
* They attended the breast feeding clinic complaining from insufficiency of lactation within the 1st month after normal vaginal delivery and they were using mixed feeding (Both breast and bottle feeding at least 3 bottles per day and not more than 6 bottles).
* They had approximately the same nutrition as well as, education level

Exclusion Criteria:

* lactating mothers who suffered from post-partum hemorrhage
* cardio respiratory disease
* diabetes mellitus
* breast cancer
* previous surgeries in the chest, breast or the surrounding area
* anemia
* those who had any causes that hindering their normal breast feeding as (retraced, cracked, inflamed or inverted nipples)
* Women receiving contraceptive pills,
* conditions related to the infant that affect the lactation process were excluded such as congenital conditions of infant mouth: tongue tie, cleft of the soft palate and congenital heart disease of the infant

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
serum prolactin | 12 weeks after treatment
  the mean difference in the value of serum prolactin between the three studied groups measured at post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maged AM, Hassanin ME, Kamal WM, Abbassy AH, Alalfy M, Askalani AN, El-Lithy A, Nabil M, Farouk D, Hussein EA, Hammad B. Effect of Low-Level Laser Therapy versus Electroacupuncture on Postnatal Scanty Milk Secretion: A Randomized Controlled Trial. Am J Perinatol. 2020 Oct;37(12):1243-1249. doi: 10.1055/s-0039-1693428. Epub 2019 Jul 21. PMID 31327162